CLINICAL TRIAL: NCT06972706
Title: Efficacy and Safety of Shatavari in Women Sexual Wellness: A Prospective, Randomized, Double-Blind, Three-arm, Parallel, Placebo-Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SF Research Institute, Inc. (Network)
Collaborators: Ixoreal Biomed Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SHT-1077-2024-02
Record Dates: First submitted 2024-11-29; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-11

CONDITIONS: Sexual Health
MeSH Terms: interventions — Ashwagandha

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Shatavari (Experimental): One capsule of Shatavari 300 mg (contains Shatavari extract) once a day, orally with water.
  Interventions: Dietary Supplement: Shatavari
- Shatavari + Ashwagandha (Experimental): One capsule of Shatavari (300mg) + Ashwagandha (250mg) (contains Shatavari + Ashwagandha root extract) once a day, orally with water.
  Interventions: Dietary Supplement: Shatavari + Ashwagandha extract
- Placebo (Placebo Comparator): One capsule of Placebo 300 mg (contains starch extract) once a day, orally with water.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Shatavari — Shatavari is scientifically known as Asparagus racemosus. One capsule containing Shatavari 300mg should be taken once daily.
  Arms: Shatavari
Dietary Supplement: Shatavari + Ashwagandha extract — Shatavari is scientifically known as Asparagus racemosus along with Ashwagandha root extract scientifically known as Withania somnifera. One capsule containing Shatavari 300mg + Ashwagandha root extract 250mg should be taken once daily.
  Arms: Shatavari + Ashwagandha
Dietary Supplement: Placebo — Placebo (starch)
  Arms: Placebo

SUMMARY:
This is a Multi-center, Multi-national, Prospective, Randomized, Double-Blind, Placebo- Controlled three arm study to evaluate the efficacy and safety of Shatavari in Women Sexual Wellness. Participants will be randomized to either one of the three treatment arms.Participants will then be asked to either take one capsule containing Shatavari or Shatavari + Ashwagandha or Placebo orally once daily in the morning after breakfast with a glass of water for 8 weeks. All the subjects will be asked to continue their routine diet and physical activities during the whole study period. The primary objective is to assess the efficacy of Shatavari capsules for improvement in Women Sexual Wellness. The secondary objective is to assess the safety of Shatavari capsules in healthy women.

DETAILED DESCRIPTION:
To qualify for the study, participants must be Women between 18 to 55 years of age. Women must be willing to have 4 or more attempts of sexual intercourse each month. Women presenting with signs and symptoms suggestive of stress (e.g., difficulty, concentrating, physical exhaustion, anxiety, restlessness, insomnia, headache, fatigue, loss of appetite, worry, sweating, mental confusion, etc.) are enrolled.

In this study, a maximum of 51 patients will be enrolled and the goal is to complete the study with at least 45 patients.

After signing this consent form, participants will answer questions regarding their medical history, including any medications they are taking. Physical exams with vital signs (pulse, temperature, sitting blood pressure and respiratory rate) will be performed at both visits by a professional trained to perform this testing. It may be a Nurse (RN or LPN), Phlebotomist, or Medical Doctor.

A blood sample will be required from subjects. Subject's right or left arm will be used as the blood draw site, requiring a 5mL sample. The blood will be analyzing Sr. Estradiol, FSH, LH, Testosterone levels. These blood draws will be administered by a professional trained to perform this testing. It may be a Nurse (RN or LPN), Phlebotomist or Medical Doctor.

All eligible participants, will be given the required quantity of the study medication for self-administration, sufficient till the Visit 3- End of study visit, 8 weeks ± 4 Days. Participants will be randomized to either one of the three treatment arms.

Participants will be instructed to take one capsule of study medication to which they are randomized after breakfast, with ambient temperature water for 8 weeks at home. Participants will be asked to visit the site for Visit 2 (4 weeks ± 4 Days), Visit 3 (8 weeks ± 4 Days). Adverse events and concomitant medication will be recorded throughout the study. Participants will be asked to get used and unused study medications and their subject diaries in this visit. All the participants will be asked to continue their routine diet and physical activities during the whole study period.

The primary end point is the mean change in scores for Female Sexual Function Index (FSFI) from baseline. And the secondary end points are mean changes scores for Satisfying Sexual Events (SSEs), Female Sexual Distress Scale (FSDS), Profile of Mood States, Oxford Happiness Questionnaire (OHQ), Pittsburgh Sleep Quality Index (PSQI) Questionnaire and mean changes in Serum hormones (Sr. Estradiol, FSH, LH, Testosterone) levels from baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Women between 18 to 55 years of age.
2. Women willing to have 4 or more attempts of sexual intercourse each month.
3. Women presenting with signs and symptoms suggestive of stress (e.g., difficulty, concentrating, physical exhaustion, anxiety, restlessness, insomnia, headache, fatigue, loss of appetite, worry, sweating, mental confusion, etc.).
4. Participants who are reliable, honest, compliant, and agree to co-operate with all trial evaluations as well as to be able to perform them as per investigator's opinion.
5. Participants having sufficient understanding to communicate effectively with the investigator and are willing to discuss their sexual functioning with the investigative staff.
6. Able to read and write in English or any other vernacular language.
7. No plan to commence new treatments over the study period.
8. Must have the ability and willingness to sign an informed consent and to comply with all study procedures

Exclusion Criteria:

1. Participants taking any form of herbal extract in the last 3 months before study entry.
2. Participants who are on hormone replacement therapy (HRT) for more than 3 months.
3. Participants with any active medical, surgical, or gynaecological problems.
4. Participants with a history of alcohol, tobacco dependence, or any other substance abuse
5. Participants with clinically relevant cardiovascular, gastrointestinal, hepatic, neurologic, endocrine, haematologic or other major systemic diseases making implementation of the protocol or other interpretation of the study result difficult.
6. Participants with mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
7. Participants with evidence of uncooperative attitude, including poor compliance.
8. Participants with inability to attend follow-up visits.
9. Patients with known hypersensitivity to Shatavari, Ashwagandha or any of the ingredients of study medication.
10. Patients who had participated in other clinical trials during the previous 3 months.
11. Patients who have any clinical condition, according to the investigator who does not allow safe fulfilment of clinical trial protocol.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2024-10-26 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Female Sexual Function Index (FSFI) | FSFI assessment will be done at Visit 1, Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1), Visit 2 (Week 4), and Visit 3- End of study visit, (Week 8).
  FSFI questions are coded from 0.0 to 5.0. Based on clinical considerations, the scale is considered to have six sexual domains: desire, arousal, lubrication, orgasm, satisfaction, pain. Each domain is contributing to the overarching construct of female sexual function. The maximum score for each domain is 6.0, obtained by summing item responses and multiplying by a correction factor. The total composite sexual function score is a sum of domain scores and ranges from 2.0 (not sexually active and no desire) to 36.0.

SECONDARY OUTCOMES:
Satisfying Sexual Events (SSEs) | SSEs assessment will be done at Visit 1, Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1), Visit 2 (Week 4), and Visit 3- End of study visit, (Week 8).
  SSE included subject's inputs for number of intercourse and non-intercourse sexual events, number of orgasms, level of sexual desire, and satisfying sexual activity experienced. The subjects will be asked to mark a score for their sexual desire. They will be asked, "Indicate your most intense level of sexual desire in the last 24 hours/since your last visit." Potential responses included "no," "low," "moderate," or "strong", scored 0-3 (0 indicating no desire and 3 indicating the highest level of desire)
Female Sexual Distress Scale (FSDS) | FSDS assessments will be done at Visit 1, Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1), Visit 2 (Week 4), and Visit 3- End of study visit, (Week 8).
  The Female Sexual Distress Scale (FSDS), a 12-item patient-reported outcome (PRO) instrument, was developed to measure sexually related personal distress in women. Both the original 12-item version and the 13-item FSDS-Revised (FSDS-R) version have been shown to have a high degree of internal consistency, test-retest reliability, and discriminative validity to distinguish between sexual function and dysfunction among women.
  The FSDS-R psychometric instrument with a 7-day recall demonstrated good discriminant validity, high test-retest reliability, and a high degree of internal consistency in measuring sexually related personal distress in women
Profile of Mood States (POMS, abbreviated version) | POMS assessment will be done at Visit 1, Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1), Visit 2 (Week 4), Visit 3 End of study visit, (Week 8).
  The POMS is a 40-item questionnaire rated on a 5-point Likert Scale, asking respondents how they feel right now. Scores are calculated for Tension, Anger, Fatigue, Depression, Esteem- related affect, Vigor, Confusion, and Total Mood Disturbance.
Oxford Happiness Questionnaire (OHQ) | OHQ assessment will be done at Visit 1 (Screening Visit/ Enrolment Visit/ Baseline Visit- Day 1), Visit 2 (Week 4), and Visit 3 (Week 8).
Pittsburgh Sleep Quality Index (PSQI) | PSQI assessment will be done at Visit 1, Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1), Visit 2 (Week 4), and Visit 3 (Week 8)
  The Pittsburgh Sleep Quality Index (PSQI) is an effective instrument used to measure the quality and patterns of sleep-in adults. It differentiates "poor" from "good" sleep quality by measuring seven areas (components): subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction over the last month.
Serum Hormones | Time Frame: Blood samples for Serum hormones (Sr. Estradiol, FSH, LH, Testosterone) will be collected at Screening Visit/ Enrolment Visit/ Baseline Visit, (Day 1) and Visit 3- (Week 8)]

CONTACTS AND LOCATIONS:
Locations (1):
- San Francisco Research Institute, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided